CLINICAL TRIAL: NCT01749527
Title: Does Patient Activity Level Affect 24-Hour Pad Test Results in Stress-Incontinent Women?
Brief Title: Does Patient Activity Level Affect 24-Hour Pad Test Results in Stress-Incontinent Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St George Hospital, Australia (Other)
Responsible Party: Principal Investigator, Emmanuel Karantanis, Doctor, St George Hospital, Australia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Activity Study
Record Dates: First submitted 2012-12-11; First posted 2012-12-13 (Estimated); Last update posted 2012-12-13 (Estimated); Status verified 2012-12

CONDITIONS: 24-hour Pad Test Weight Gain With and Without Activity
Keywords: 24-hour pad test; Activity; Stress urinary incontinence
MeSH Terms: conditions — Motor Activity; Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 24-hour pad test (Other): decreased activity
  Interventions: Behavioral: minimal activity

INTERVENTIONS:
Behavioral: minimal activity — Pad test with minimal activity

SUMMARY:
We hypothesised that in women with stress urinary incontinence, the severity of leakage on a 24 hour pad test was affected by activity.

DETAILED DESCRIPTION:
We asked women to perform two separate pad tests, one with normal activity, and another with decreased activity.

ELIGIBILITY:
Inclusion Criteria:

* Stress urinary incontinence

Exclusion Criteria:

* language other than english

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-03; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
24-hour pad test weight gain (mls) | 24 hours